CLINICAL TRIAL: NCT00253305
Title: Phase IIB Efficacy and Safety Study of Four Topical Gel Formulations of Anti-Fungal Agents, MQX-5858, MQX-5859, MQX-5866, and MQX-5867, Versus Vehicle in the Treatment of Tinea Unguium.
Brief Title: Topical Gel Anti-Fungal Agent for Tinea Unguium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MQT-05-001
Record Dates: First submitted 2005-11-13; First posted 2005-11-15 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Onychomycosis
Keywords: tinea unguium; onychomycosis
MeSH Terms: conditions — Onychomycosis

INTERVENTIONS:
Drug: Organogel of naftifine, 2%
Drug: Organogel of terbinafine, 2%
Drug: Organogel of naftifine, 6%
Drug: Organogel of terbinafine, 6%

SUMMARY:
The purpose of this study is to compare, in a controlled fashion, the response to two anti-fungal agents, naftifine or terbinafine, with vehicle in novel topical gel formulations in the treatment of subjects with distal subungual tinea unguium of the toenails (onychomycosis).

The formulation used as the vehicle for the active agents has been shown in earlier studies to facilitate the penetration of the active agent through fungally-infected nails. This study will examine dose-response and agent differences in terms of efficacy and safety.

Once the subject has qualified for the study, he/she will be randomly assigned to one of five study groups, dispensed appropriate study medication and instructed to apply one drop to the great toe designated for study.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of distal subungual tinuea unguium of one great toenail.
* between 20 - 65% infected area for target nail
* 2 mm of clear nail proximally on target nail
* positive dermatophyte culture and positive KOH test
* able to sign informed consent
* understand requirements of study
* females must be post-menopausal or agree to use approved contraceptives throughout the study

Exclusion Criteria:

* patients with nails infected with organisms other than dermatophytes
* patients with proximal subungual tinea unguium
* patients with spikes of disease extending to nail matrix
* patients with more than 5 infected nails
* patients with confounding problems/ abnormalities of target nail
* patients with screening lab values more than 20% of normal
* patients with known hypersensitivity to test material components
* patients requiring systemic medications that may interfere with study
* patients with a poor history of compliance with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-09

PRIMARY OUTCOMES:
Quanitative improvement in toenail appearance.
Assessment of dermatophyte culture and KOH examination.
Frequency and severity of adverse events.

SECONDARY OUTCOMES:
Time to achieve 90% and 100% clearance of fungus from nail.
Assessment of treatment success.
Assessment of mycological success.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Greater Miami Skin and Laser Center, Miami Beach, Florida
  - Washington University, St Louis, Missouri
  - Northwest Cutaneous research, Portland, Oregon